CLINICAL TRIAL: NCT04620902
Title: Detection of AD Biomarkers in Tear Fluid
Acronym: SmartTears
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-4-100
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Dementia: Dementia
  Interventions: Other: Tear sampling
- MCI: Mild cognitive impairment
  Interventions: Other: Tear sampling
- SCD: Subjective cognitive decline
  Interventions: Other: Tear sampling
- HC: Cognitively healthy control
  Interventions: Other: Tear sampling

INTERVENTIONS:
Other: Tear sampling — Tear sampling using Schirmer's strips

SUMMARY:
Detection of AD biomarkers in tear fluid

ELIGIBILITY:
Inclusion Criteria:

* . Inclusion criteria were an MMSE score ≥ 20 and a CDR score from 0 to 1, thereby including patients across the whole clinical spectrum (i.e. from subjective cognitive disorder to (mild) dementia).

Exclusion Criteria:

* Exclusion criteria at baseline were neurological diseases (such as Normal Pressure Hydrocephalus, Morbus Huntington, brain tumor, epilepsy, encephalitis, recent Transient Ischemic Attack (TIA) or cerebrovascular accident (CVA) (< 2 years), or TIA/CVA with concurrent (within three months) cognitive decline) and a history of psychiatric disorders (such as schizophrenia, bipolar disorder or psychotic problems, current major depressive disorder (within 12 months), or alcohol abuse).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 60 patients and nine cognitively healthy age-matched controls (HC) were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Level of AD biomarkers in tear fluid | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Hospital Maastricht, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided